CLINICAL TRIAL: NCT01075529
Title: Model for Early Prediction of Clinical Response in Patients With Major Depression Receiving Fluoxetine
Brief Title: Early Prediction of Fluoxetine Response
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kaohsiung Kai-Suan Psychiatric Hospital (Other Government)
Responsible Party: Ching-Hua Lin, M.D., Kaohsiung Kai-Suan Psychiatric Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KSPH-2007-16
Record Dates: First submitted 2010-02-24; First posted 2010-02-25 (Estimated); Last update posted 2010-02-25 (Estimated); Status verified 2010-02

CONDITIONS: Major Depressive Disorder
Keywords: major depressive disorder, fluoxetine, Hamilton Rating Scale for Depression (HAM-D-17)
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Fluoxetine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- fluoxetine (No Intervention)
  Interventions: Drug: fluoxetine

INTERVENTIONS:
Drug: fluoxetine — fluoxetine 20 mg/d

SUMMARY:
The purpose of this study is to identify what degree of symptom changes during the early weeks could be used to predict eventual nonresponse at week 6 among depressive inpatients taking fluoxetine.

DETAILED DESCRIPTION:
Patients with major depressive disorder will receive 20 mg/day of fluoxetine for six weeks. Symptom severity was assessed by the 17-item Hamilton Depression Rating Scale (HAMD-17) at weeks 0, 1, 2, 3, 4 and 6. Stable response is defined as a reduction of 50% or more of the HAMD-17 score at week 4 and week 6 of treatment. Receiver operating characteristic curve will be used to determine the cutoff point of the percentage of HAMD-17 score reduction between stable responders and nonresponders at weeks 1, 2, 3 and 4.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of major depressive disorder
* HAM-D-17 ≧17
* written informed consent

Exclusion Criteria:

* Comorbid of substance abuse/dependence
* Comorbid with mental disorders due to general medical conditions
* Past history of treatment-resistant depression
* Severe physical problems
* pregnant women
* lactation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2007-03; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Stable response was defined as a reduction of 50% or more of the HAMD-17 score at week 4 and week 6 of treatment | 6 weeks after initiation of fluxetine

SECONDARY OUTCOMES:
CGI, GAF, Zung's Depression Scale, Short-Form 36, auditory evoked potential, psychomotor speed | 6 weeks after initiation of fluxetine

CONTACTS AND LOCATIONS:
Overall Officials: Ching-Hua Lin, M.D., Principal Investigator — Kai-Suan Psychiatric Hospital
Locations (1):
- Kai-Suan Psychiatric Hospital, Kaohsiung City, Taiwan

REFERENCES:
- [Result] Tollefson GD, Holman SL. How long to onset of antidepressant action: a meta-analysis of patients treated with fluoxetine or placebo. Int Clin Psychopharmacol. 1994 Winter;9(4):245-50. doi: 10.1097/00004850-199400940-00003. PMID 7868846
- [Result] Bech P. Meta-analysis of placebo-controlled trials with mirtazapine using the core items of the Hamilton Depression Scale as evidence of a pure antidepressive effect in the short-term treatment of major depression. Int J Neuropsychopharmacol. 2001 Dec;4(4):337-45. doi: 10.1017/S1461145701002565. PMID 11806859
- [Result] Katz MM, Tekell JL, Bowden CL, Brannan S, Houston JP, Berman N, Frazer A. Onset and early behavioral effects of pharmacologically different antidepressants and placebo in depression. Neuropsychopharmacology. 2004 Mar;29(3):566-79. doi: 10.1038/sj.npp.1300341. PMID 14627997
- [Result] Farabaugh A, Mischoulon D, Fava M, Wu SL, Mascarini A, Tossani E, Alpert JE. The relationship between early changes in the HAMD-17 anxiety/somatization factor items and treatment outcome among depressed outpatients. Int Clin Psychopharmacol. 2005 Mar;20(2):87-91. doi: 10.1097/00004850-200503000-00004. PMID 15729083
- [Result] Trivedi MH, Morris DW, Grannemann BD, Mahadi S. Symptom clusters as predictors of late response to antidepressant treatment. J Clin Psychiatry. 2005 Aug;66(8):1064-70. doi: 10.4088/jcp.v66n0816. PMID 16086624
- [Derived] Yang WC, Lin CH, Wang FC, Lu MJ. Factors related to the improvement in quality of life for depressed inpatients treated with fluoxetine. BMC Psychiatry. 2017 Aug 25;17(1):309. doi: 10.1186/s12888-017-1471-3. PMID 28841824